CLINICAL TRIAL: NCT04829227
Title: Safety and Efficacy of Sofwave Treatment to Lift Lax Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Sofwave05
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2021-03

CONDITIONS: Skin Laxity
Keywords: Laxity Brow Lifting Skin Saggy
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- face and/or neck and/or submental zones (Experimental): the full face and/or neck and/or submental zones including 1. -The forehead and temples (left and right including the peri orbital zone) to lift the eyebrows 2. The cheeks (left and right including perioral zone and nasolabial folds) 3. Submental and sides of the neck
  Interventions: Device: Sofwave
- "off the face" areas (Experimental): "off the face" areas: abdomen, or arms or thighs or Décolleté.
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.

SUMMARY:
Open-label, non-randomized 2 arms prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
This study is a two-arm study. Eligible patients will receive 2-4 face and/or neck and/or submental or "off the face" (abdomen, or arms, or thighs, or Décolleté) treatments (per PI discretion, 2-12 weeks apart) using the Sofwave System. In arm 1, each investigational site would treat the full face and/or neck and/or submental zones including 1. -The forehead and temples (left and right including the peri orbital zone) to lift the eyebrows 2. The cheeks (left and right including perioral zone and nasolabial folds) 3. Submental and sides of the neck (left and right) to lift lax skin. In arm 2, each site would treat "off the face" areas: abdomen, or arms or thighs or Décolleté. Each patient could be assigned to both arms. Treatment may be administered after the enrollment and screening at the first visit or it may occur at a later date following the enrollment and screening activities based on site scheduling availabilities. All patients will return to the clinic for one follow up visitat3 months ± 2 weeks post last treatment (FU1) and a second optional visit at 2. 6 months ± 2 weeks post last treatment (FU2; optional). Each treatment visit will also serve as a follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 35-80.
2. Non-Smoker.
3. Fitzpatrick skin type I-VI.
4. Desire to lift lax skin in the neck and submental and/or to lift the brows.
5. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent
7. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Presence of any active systemic or local infections.
3. Presence of active local skin disease that may alter wound healing.
4. Severe solar elastosis.
5. History of smoking in past 10 years.
6. History of chronic drug or alcohol abuse.
7. Excessive subcutaneous fat on the cheeks.
8. Significant scarring in the area to be treated.
9. Severe or cystic facial acne, acutance uses during past 6 months.
10. Presence of a metal stent or implant in the facial area (dental implants and/or braces are not excluded).
11. Inability to understand the protocol or to give informed consent.
12. History of cosmetic treatments in the facial area to be treated, including facial skin-tightening procedure within the 6 months ; injectable (Botox or fillers) of any type within the 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift, blepharoplasty, or brow lift (including contour threads) within the past 12 months.
13. Taking Isotretinoin or other oral retinoid within the past 6 months; taking anti-platelet or anti-coagulant within the past 2 weeks.
14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Improvements in lifting of lax tissue | 3 and 6 months post last treatment
  as assessed by independent masked evaluators of pre and post treatment images.

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Amir, MD, Study Director — Sofwave
Locations (4):
- United States (4):
  - SLSS, a Division of Schweiger Dermatology Group Research Office, Hackensack, New Jersey
  - The Practice of Brian S. Biesman, MD, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - McDaniel Institute of Aging Research, Virginia Beach, Virginia